CLINICAL TRIAL: NCT04086433
Title: Gastric Tissue Stapler Comparison Study
Status: Completed | Type: Observational
Sponsor: Standard Bariatrics (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-2018-01
Record Dates: First submitted 2019-07-29; First posted 2019-09-11 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Gastric Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Arm A - Echelon Stapler: Excised gastric tissue specimens will be resected with the Echelon Stapler (Ethicon, size: 60mm, "Echelon") and evaluated for burst pressure and staple malformation
  Interventions: Device: gastric tissue resection
- Arm B - Titan Stapler: Excised gastric tissue specimens will be resected with the Titan SGS Stapler (Standard Bariatrics, "Titan") and evaluated for burst pressure and staple malformation
  Interventions: Device: gastric tissue resection

INTERVENTIONS:
Device: gastric tissue resection — human stomach specimens will be resected with the surgical staplers for pressure testing and staple malformation assessment

SUMMARY:
This study is conducted to compare performance characteristics of staple lines resecting the stomach in excised human gastric tissue with existing Echelon Flex Powered Plus GST System (Ethicon, size: 60mm, "Echelon") stapler and the Titan SGS (Standard Bariatrics, "Titan").

The Study is a single center clinical trial, randomized (1:1, Arm A - Ethicon Echelon 60 application, Arm B - Standard Bariatrics Titan SGS application) which utilizes the excised stomach tissue from up to 75 adults undergoing laparoscopic sleeve gastrectomy (LSG). This study will be conducted in the USA.

ELIGIBILITY:
Inclusion Criteria:

1. Laparoscopic sleeve gastrectomy patients at study site, ages 18 to 80

Exclusion Criteria:

1. Prior gastric surgery (lap band, Nissen fundoplication, G tube, greater curve plication, etc.)
2. Gastric lesion recognized during surgery (entire specimen would be sent to pathology)
3. Stomach damaged during extraction

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing Laparoscopic Sleeve Gastrectomy
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Hoffman, MD, FACS, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Echelon Stapler | Arm B - Titan Stapler
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Echelon Stapler | Arm B - Titan Stapler | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 41 [28 to 57] | 46 [19 to 66] | 44 [19 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pressure Evaluation
Description: Burst pressure will be assessed in the specimen with one staple line (i.e. the test staple line) with a pressure volume curve recorded.
Time Frame: immediately post operative
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Arm A - Echelon Stapler | Arm B - Titan Stapler
Number analyzed (Participants) | 17 | 18
mmHg | 126 [46 to 226] | 163 [82 to 259]

2. Primary Outcome: Staple Malformation
Description: Staple line specimen will be sent to an independent laboratory for imaging. Percentage of malformed staples in test staple line will be recorded by an independent assessor.
Time Frame: through study completion, anticipate within 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Not applicable. Investigation performed on excised tissue.
Description: Not applicable. Investigation performed on excised tissue.
Arm/Group | Arm A - Echelon Stapler | Arm B - Titan Stapler
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Echelon Stapler (N=0) | Arm B - Titan Stapler (N=0)
Other (Product Issues) | 0 | 0 — All-cause mortality, serious and other adverse events were not monitored assessed. These are not applicable to this study because the study was performed on previously excised tissue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04086433/Prot_000.pdf